CLINICAL TRIAL: NCT04212338
Title: Effect of Music Intervention on Pain, Anxiety, Physiological Variables, Patient Satisfaction, and Surgeon-Patient Cooperation in Intravitreal Injection
Brief Title: Effect of Music Intervention on Intravitreal Injection
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Afyonkarahisar Health Sciences University (Other)
Responsible Party: Principal Investigator, Yeliz Ciğerci, Director, Afyonkarahisar Health Sciences University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: 2019/76
Record Dates: First submitted 2019-12-24; First posted 2019-12-27 (Actual); Last update posted 2019-12-27 (Actual); Status verified 2019-12

CONDITIONS: Music Intervention

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- study group 1 (Experimental): Before intravitreal injection music intervention: These patients received the standard treatment and listened to music for a period of 15 minutes 30 minutes before the injection.
  Interventions: Other: Before intravitreal injection music intervention
- study group 2 (Experimental): During-intravitreal injection music intervention:These patients received the standard treatment and listened to music during the injection (approximately 5 minutes).
  Interventions: Other: during intravitreal injection music intervention
- control group (No Intervention): The music intervention was not conducted with the patients in the control group. These patients received the standard treatment.

INTERVENTIONS:
Other: Before intravitreal injection music intervention — The patients in the Before-IVTI group listened to music for a period of 15 minutes 30 minutes before the injection.
  Arms: study group 1
Other: during intravitreal injection music intervention — The patients in the During-IVTI group listened to music during the injection (approximately 5 minutes).
  Arms: study group 2

SUMMARY:
The objective of this study was to examine the effect of music intervention in the before-intravitreal injection (IVTI) and during-IVTI periods on patients' anxiety, the sensation of pain, physiological variables, satisfaction, and surgeon-patient cooperation. The study used a randomized controlled experimental design. The study was conducted with a total of three groups: two experimental (Before-IVTI (Group1) and During-IVTI music intervention group (Group 2)) and one control group. Each of the experimental and control groups consisted of 75 patients. The patients' anxiety was evaluated using the VAS anxiety scale, pain using the VAS pain scale; surgeon-patient cooperation using the Numeric Rating Scale; and patient satisfaction with a 5-point likert-type satisfaction scale.

ELIGIBILITY:
Inclusion Criteria:

* The participants were patients aged 18 or above,
* Who did not have a hearing/speech impairment, a mental problem or a diagnosed psychiatric disorder, who had not received a diagnosis of depression, who volunteered to participate in the study, and on whom elective IVTI was carried out, or who had undergone IVTI previously.

Exclusion Criteria:

* The participants were patients aged under 18 years
* Who had a hearing/speech impairment, a mental problem or a diagnosed psychiatric disorder, who had received a diagnosis of depression, who did not volunteered to participate in the study, and or who had not undergone IVTI previously.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 219 (Actual)
Dates: Start 2019-03-11 (Actual); Primary Completion 2019-05-24 (Actual); Study Completion 2019-05-24 (Actual)

PRIMARY OUTCOMES:
Visual Analog Scale for Anxiety (VAS-A) | 1 day
  VAS-A is a measurement tool, in which 0 represents feeling "no anxiety" while 10 represents "I feel extremely anxious".29 An increase in score indicates an increase in the anxiety experienced by the patient. This indicates that VAS-A is a reliable and accurate measurement tool despite its brevity. The VAS-A scale was applied to patients before, immediately after, and 15 minutes after the injection.

SECONDARY OUTCOMES:
Visual Analog Scale for Pain (VAS) | 1 day
  VAS scale is a single-dimensional scale that is commonly used to evaluate pain severity. According to the VAS, pain severity is rated from 0 (no pain) to 10 (the greatest imaginable pain). Any score under 3 on the scale is considered "mild pain", scores between 3 and 6 are "moderate pain" and any score above 6 is "severe pain". The VAS was applied both immediately after the injection and 15 minutes afterwards in order to determine the severity of the pain that the patients felt during the injection.

OTHER OUTCOMES:
Surgeon-patient cooperation | 1 day
  Numeric Rating Scale (NRS) was used. This scale allows for a score of between 0 and 10 points.A score of 0 indicates that the patient was totally noncompliant with the surgeon's instructions and a score of 10 indicates that the patient was totally compliant. The NRS was used by the surgeon for each patient immediately after the conclusion of the injection.
Patient Satisfaction | 1 day
  In this study, on the basis of the review of the literature, satisfaction was evaluated using a 5-point Likert-type scale. The patients were asked to respond "Very Unsatisfied", "Unsatisfied", "Neutral", "Satisfied", or "Very Satisfied". The patients' levels of satisfaction were evaluated 15 minutes after the injection.

CONTACTS AND LOCATIONS:
Overall Officials: Yeliz Ciğerci, Principal Investigator — +90 272 444 0304
Locations (1):
- Afyonkarahisar Health Science University, Afyonkarahisar, Centre, Turkey (Türkiye)